CLINICAL TRIAL: NCT00643318
Title: A Prospective Evaluation of Outcomes of Radiosurgical Treatment of Early Stage Non-Small Cell Lung Cancer (NSCLC)
Brief Title: CyberKnife Radiosurgical Treatment of Inoperable Early Stage Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Accuray Incorporated (Industry)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCL001.0
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2019-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer; lung tumor; non-small cell lung cancer; NSCLC; CyberKnife; radiosurgery; lung surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiosurgery; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CyberKnife Stereotactic Radiosurgery (Experimental)
  Interventions: Radiation: CyberKnife Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: CyberKnife Stereotactic Radiosurgery — Central tumors defined as < 2 cm from carina and < 2 cm from right and left mainstem bronchus and/or < 2 cms from the right and left upper lobe bronchus, bronchus intermedius, middle lobe bronchus, and the right and left lower lobe bronchus. For central tumors, 4 fractions of 12 Gy will be delivered (12 Gy x 4 fractions = 48 Gy)
  Peripheral tumors are defined as being > 2 cms from the carina and > 2 cms from the right and left mainstem bronchus and/or > 2 cms from the right and left upper lobe bronchus, bronchus intermedius, middle lobe bronchus and the right and left lower lobe bronchus. For peripheral tumors, 3 fractions of 20 Gy will be delivered (20 Gy x 3 fractions = 60 Gy)
  Other Names: CyberKnife; Stereotactic Radiosurgery; Radiosurgery; Radiation Therapy

SUMMARY:
The purpose of this study is to assess the short and long-term outcomes after CyberKnife stereotactic radiosurgery for early stage non-small cell lung cancer (NSCLC) in patients who are medically inoperable.

DETAILED DESCRIPTION:
The objectives of this clinical evaluation are to assess the outcomes of patients who undergo stereotactic radiosurgery (SRS) to treat primary early stage non-small cell lung cancer (NSCLC) in patients (comprising of two cohorts, peripheral and central) who are not candidates for surgical resection because of high operative risks. In particular, the effect of CyberKnife SRS on clinical response rate, local control, progression-free survival, overall survival, dyspnea and QOL (for U.S. sites), and radiological findings over two years after treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be over the age of 18 years
2. Pulmonary nodule with maximum diameter ≤ 5 cm
3. Histological confirmation of primary NSCLC
4. The following stage of NSCLC patients are eligible:

   * Stage I: T1 N0 M0 or T2 N0 M0 (Tumor size ≤ 5 cm)
   * Stage II: T3 N0 M0 (Chest wall invasion only, Tumor size ≤ 5 cm)
5. ECOG/Zubrod status of 0, 1 or 2
6. Thoracic surgery consultation should be obtained from a Board Certified Thoracic surgeon who in collaboration with a radiation oncologist should determine that the patient is not a surgical candidate.
7. In order to be considered medically inoperable, the patient must meet at least one major criteria or a minimum of 2 minor criteria as described below:

   MAJOR CRITERIA:
   1. FEV1 < 50% or predicted postoperative FEV1 < 40%
   2. DLCO < 50% or predicted postoperative DLCO < 40%
   3. Exercise induced maximal exercise oxygen consumption M VO2 < 15 mL/kg/min
   4. High-risk cardiac disease: Any one of the following:

      * Poor left ventricular function (defined as an ejection fraction of <=20%)
      * Unstable coronary syndromes (unstable angina or severe angina Canadian class III or IV).
      * Severe valvular disease (critical valvular stenosis),
      * Recent myocardial infarction (< 1 month),
      * Significant arrhythmia defined by one of the following: High-grade AV block, Symptomatic ventricular arrhythmias in the presence of underlying heart disease, Supraventricular arrhythmias with uncontrolled ventricular rate

   MINOR CRITERIA:
   1. Age > 75
   2. Pulmonary hypertension (defined as a pulmonary artery systolic pressure greater than 40 mm Hg)
   3. Oxygen requirement (using the Medicare criteria for home oxygen requirements [i.e., room air oxygen saturation of 88% or less])
   4. Resting or exercise arterial pO2 ≤ 55 mm Hg OR SpO2 ≤ 88%.
   5. pCO2 > 45 mm Hg
   6. Congestive heart failure (any three of the following must be documented: dyspnea, peripheral edema, chest x-ray with interstitial edema or cardiomegaly, rales, or congestion)
   7. Moderately depressed left ventricular function (defined as an ejection fraction of 21-40% or less)
   8. Severe cerebral (with CVA or recent TIA) or severe peripheral vascular disease
   9. Diabetes Mellitus with severe organ damage such as ESRD, Blindness, Vascular disease.
   10. Severe end organ damage from other causes resulting in ESRD, cirrhosis of the liver or vascular disease
   11. FEV1 51%-60% or predicted postoperative FEV1 41-50%
   12. DLCO 51-60% or predicted postoperative DLCO 41-50%
   13. Modified Medical Research Council Dyspnea Scale ≥ grade 3
8. Females of child-bearing age must be using a reliable form of birth control.
9. The patient must have a PET-CT scan within 8 weeks of registration.
10. The patient must provide a signed and dated written informed consent PRIOR to registration and prior to undergoing any study-related procedures.
11. The patient must provide written authorization to allow the use and disclosure of their protected health information.

Exclusion Criteria:

1. Excluding the primary cancer targeted for this treatment, the patient has a prior history of cancer (within the last 5 years) or concurrent cancer other than basal cell or squamous skin cancer.
2. Visible endobronchial lesion seen in the trachea, carina, major bronchus, lobar or segmental bronchus on bronchoscopy or microscopic disease detected in the trachea, carina, major bronchus, lobar or segmental bronchus.
3. The patient's weight exceeds the tolerances of the institution's imaging and CyberKnife platform/couch.
4. The patient has received thoracic radiation therapy in the same field as the planned treatment area in the past.
5. The patient has completed chemotherapy within less than 30 days of treatment.
6. T2: Tumor size > 5 cm, T3 tumors (except T3 by virtue of chest wall invasion and ≤ 5 cm), T4 tumors. Presence of N1, N2 or N3 disease per previously described criteria would be excluded.
7. Pancoast tumors would be excluded.
8. Current distant metastatic disease (M1) (preferably biopsy proven).
9. The patient is a female with child-bearing potential who refuses to take a pregnancy test prior to treatment.
10. The patient is pregnant or a female who is nursing an infant.
11. The patient is planning on undergoing systemic therapy within 2 weeks after the last fraction of radiation
12. The patient has an active systemic or pulmonary infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Local progression-free survival, local disease progression, clinical response rate, regional recurrence-free survival, distant recurrence-free survival. | 5 years

SECONDARY OUTCOMES:
To characterize and compare quality of life before and after stereotactic radiosurgery treatment. To assess procedure-related outcomes after stereotactic radiosurgery of lung tumors. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: James Luketich, MD, Study Chair — University of Pittsburgh Medical Center
Locations (23):
- United States (21):
  - St Joseph's Hospital/Barrow Neurological Institute, Phoenix, Arizona
  - Community Regional Medical Center, Fresno, California
  - Stanford University, Palo Alto, California
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Denver CyberKnife, Lone Tree, Colorado
  - North Florida Radiation Oncology, Gainesville, Florida
  - Naples Community Hospital, Naples, Florida
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Advocate Christ Med Center, Oak Lawn, Illinois
  - Parkview Cancer Center, Fort Wayne, Indiana
  - St. Catherine's Hospital, Munster, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - St. Louis University Hospital, St Louis, Missouri
  - St. Mary's Regional Medical Center, Reno, Nevada
  - St. Anthony's Hospital, Oklahoma City, Oklahoma
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor Research Institute, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Multicare Health System, Tacoma, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- China (2):
  - Ruikang Hospital, Nanning, Guangxi
  - Tianjin Medical University Cancer Institution and Hospital, Tianjin

REFERENCES:
- See also: Accuray Website — http://www.accuray.com